CLINICAL TRIAL: NCT07087509
Title: Evaluation of the Safety and Performance of the TriOSS®: A Retrospective Observational Study in Orthopaedic Area
Acronym: TriOSSOrto01
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely due to the inability to collect retrospective clinical data within the required contractual and regulatory deadlines. Although ethical approval was obtained, data collection was not performed.
Sponsor: Bioceramed (Industry)
Collaborators: Hospital dos Lusíadas (Other)
Responsible Party: Sponsor
Other Study IDs: TriOSSOrto01
Record Dates: First submitted 2025-07-01; First posted 2025-07-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bone Defect; Orthopedic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to collect real-world clinical data to gather information on the performance and safety of the TriOSS® when used according to its intended purpose and current clinical applications. The results of the clinical study will serve as clinical evidence for the device's clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (age > 18 years old);
* Patients with osseous defects, either of trauma origin, surgically created, or associated with spinal degenerative diseases that require segmental fusion of the spine.
* Patients with bone skeletal defects that are not intrinsic to the stability of the bone structure.

Exclusion Criteria:

* Signs of local or systemic acute/ active or chronic infections;
* Metabolic affections;
* Severe degenerative diseases, conditions in which general bone grafting is not advisable;
* Implementation sites that allow product migration;
* Conditions which require structural support in the skeletal system;
* Conditions where the implantation site is unstable and not rigidly fixated;
* Sensibility to the implantable materials;
* Known hypersensitivity to the implant material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (> 18 years old) undergoing orthopaedic surgery after bone defect.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Performance Endpoint | Follow-up visits according to clinical practice and medical records: months post-surgery until a maximum of 24 months
  the success of bone consolidation on the surgery site, measured by X-ray. This includes radiological assessments (X-rays) to prove bone regeneration and assess the time required for bone consolidation.
Safety Endpoint | Follow-up visits according to clinical practice and medical records, months post-surgery, until a maximum of 24 months
  Assessment of AEs related to TriOSS® during the follow-up period of patients. Description of the event type, duration, determination of Serious Adverse Event (SAE) status, and follow-up of the adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Lusíadas Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No